CLINICAL TRIAL: NCT05816629
Title: Multiparameter Ultrasound Based-AI for the Diagnosis of Thyroid Nodules: an International Multi-center Study
Brief Title: Multiparameter Ultrasound Based-AI for the Diagnosis of Thyroid Nodules
Acronym: AI
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: Thyroid AI-2023
Record Dates: First submitted 2023-02-14; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-01

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Multiparameter ultrasound based-AI — Multiparameter ultrasound based-AI for the diagnosis of thyroid nodules

SUMMARY:
The cases that fulfill the inclusion criteria will be enrolled with written informed consent. Images and videos will be collected in accordance with the procedure, uploaded to Ruiying Cloud, followed up, and registered with basic case information, such as thyroid function, FNA/surgical pathology results, etc.

ELIGIBILITY:
Inclusion Criteria:

* 18~80 years old;
* Thyroid nodules (ACR-TI RADS category 3-5，category 3 nodules ≥1cm submitted for FNA) or clustered micro-calcifications;
* The patients schedule to perform FNA/surgery within 1 month;
* Without any history of invasive procedure of thyroid before (such as FNA,CNB, ablation, radiation, or surgery).

Exclusion Criteria:

* Incomplete data;
* Contraindications of CEUS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with thyroid nodule
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with 1827 Nodule Classification | up to 4 weeks
  nodules with Pathology or cytopathology result

CONTACTS AND LOCATIONS:
Locations (1):
- SAHZJU, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
The datasets during the current study available for participants from the sponsor on reasonable request.